CLINICAL TRIAL: NCT00373308
Title: Quality of Life Following Radical Prostatectomy
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PROS0012; 78463 (Other: Stanford University Alternate IRB Approval Number); PROS0012 (Other: Stanford University)
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will utilize the Expanded Prostate Cancer Index Composite questionnaire to learn what impact the surgery has upon the participant's sense of health, sexual and urinary quality of life.

DETAILED DESCRIPTION:
To define impact on quality of life issues for patients undergoing radical prostatectomy. This study will distribute a questionnaire to patients who are being scheduled for radical prostatectomy, both before and after surgery, to assess the impact on quality of life issues. This will provide important information regarding the temporal return of issues pertaining to quality of life.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled to undergo radical prostatectomy at Stanford

Exclusion Criteria:

- Patients treated with neoadjuvant or adjuvant hormonal therapy or radiation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo radical prostatectomy at Stanford
Sampling Method: Non-Probability Sample
Enrollment: 888 (Actual)
Dates: Start 2002-09; Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
urinary and bowel habits | before and after surgery
sexual and hormonal index as self-reported in the questionnaires | before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Chung, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No